CLINICAL TRIAL: NCT01265368
Title: A Phase 1/2, Proof-of-Principle, Multi-Center, Open-Label, Single-Arm, Non-randomized Clinical Study to Assess Safety and Efficacy of a Tumor Vaccine Consisting of Genetically Modified Allogeneic (Human) Tumor Cells for the Expression of IL-7, GM-CSF, CD80 and CD154, in Fixed Combination With a DNA-based Double Stem Loop Immunomodulator in Patients With Advanced Renal Cell Carcinoma (ASET Study)
Brief Title: A Clinical Study to Assess Safety and Efficacy of a Tumor Vaccine in Patients With Advanced Renal Cell Carcinoma (ASET)
Acronym: ASET
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mologen AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGN1601-CT1; 2009-016853-16 (EudraCT Number)
Record Dates: First submitted 2010-12-22; First posted 2010-12-23 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Stage IV Renal Cell Cancer
Keywords: Advanced Renal Cell Carcinoma; Tumor Vaccine; Cell-based Therapy
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study medication (Experimental)
  Interventions: Biological: MGN1601

INTERVENTIONS:
Biological: MGN1601 — Genetically modified allogeneic (human) tumor cells for the expression of IL-7, GM-CSF, CD80 and CD154, in fixed combination with a DNA-based double stem loop immunomodulator (dSLIM)

SUMMARY:
This is a Phase 1/2, proof-of-principle clinical study to assess safety and efficacy of a intradermally administered tumor vaccine (MGN1601). The study will be conducted in patients with advanced renal cell carcinoma.

DETAILED DESCRIPTION:
Twenty four patients with advanced RCC will be included in this open, single-arm study.

The treatment will last 12 weeks. The investigational product (MGN1601) will be administered intradermally for a total of 8 applications, whereas the first 3 applications will be administered weekly, and the following 5 applications will be administered bi-weekly.

Patients who will develop disease control (CR, PR, or SD) by week 12 will be proposed to participate in the extension phase of the study. The extension phase will be continued until disease progression in each patient, however, maximally up to week 120 (total treatment duration 2.5 years). During this time period the investigational product will be administered 5 times by weeks 24, 36, 48, 72, and 120.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 18 years of age
* Histologically confirmed renal cell carcinoma
* Radiologically confirmed advanced disease defined as unresectable locally reccurrent or metastatic disease (AJCC Stage IV)
* Previous nephrectomy
* No standard therapy is available for the patient
* At least 4 weeks after previous radiotherapy prior to study treatment
* At least 1 week after previous systemic therapy prior to study treatment
* At least one lesion measurable by modified RECIST criteria
* ECOG performance status 0-1
* Adequate organ function including hematopoietic organs
* MSKCC prognostic ctiteria < 3 predictors of short survival
* Negative urine pregnancy test in women with childbearing potential
* Women of childbearing potential and all male participants are willing to use acceptable methods of contraception (birth control pills, barriers)
* Expected adequacy of follow-up
* Signed informed consent form (ICF).

Exclusion Criteria:

* Clinically significant concomitant diseases or conditions unrelated to the underlying malignancy or therapy, which in opinion of the investigator would lead to an unacceptable risk for the subject to participate in the study
* Known hypersensitivity to any component of the study drug
* Prior or current other malignancy, except adequately treated superficial bladder cancer, basal or squamous cell carcinoma of the skin or other cancer for which the subject has been disease free for more than 3 years
* Active brain metastases except adequately treated brain metastases with no progression for at least 3 months
* Active or uncontrolled infections
* Transfusion-dependent anemia
* History of autoimmune disease or immune deficiency
* Concurrent chronic systemic immune therapy, corticosteroids or other immunosuppressant medication
* Concurrent radiotherapy within the last 4 weeks prior to study treatment and/or during the course of the study
* Concurrent immunotherapy or targeted therapy within the last 1 week prior to study treatment and/or during the course of the study
* HIV seropositivity or active hepatitis B or C infection
* Planned major surgery during the study
* Participation in other clinical studies during this clinical study
* Vaccination within 3 months prior to the first treatment day
* Any medical, mental, psychological or psychiatric condition which in opinion of the investigator would not permit the subject to complete the study or understand the patient information
* Pregnancy and/or nursing
* Presence of drug and/or alcohol abuse
* Commitment to an institution by virtue of an order issued either by judicial or administrative authorities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Assessment of safety profile of MGN1601 | Treatment phase (12 weeks), extension phase (120 weeks, if applicable), plus 5 years follow-up

SECONDARY OUTCOMES:
Assessment of potential autoimmune effects of MGN1601 | Treatment phase (12 weeks), extension phase (120 weeks, if applicable) plus 5 years follow-up (if applicable)
Assessment of the presence of MIDGE vectors | Treatment phase (12 weeks)
Assessment of the immune response to MGN1601 | Treatment phase (12 weeks), extension phase (120 weeks, if applicable)
Evaluation of clinical and radiological response to MGN1601 | Treatment phase (12 weeks), extension phase (120 weeks, if applicable) plus 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Grünwald, Prof. Dr., Principal Investigator — MHH Hannover
Locations (3):
- Germany (3):
  - Charité - Universtitäsmedizin Berlin, Klinik für Urologie, Berlin
  - Universitätsklinikum Bonn, Med. Klinik und Poliklinik, Hämatologie und Onkologie, Bonn
  - Medizinische Hochschule Hannover, Klinik für Hämatologie, Hämostaseologie, Onkologie und Stammzelltransplantation OE6860, Hanover

REFERENCES:
- See also: Related Info — http://www.mologen.com